CLINICAL TRIAL: NCT06550375
Title: Ambispective Analysis of Patient Reported Outcomes and Visual Acuity in Patients With Bilateral Implantation of Odyssey Intraocular Lenses
Brief Title: Clinical Outcomes With Bilateral Implantation of Odyssey IOLs
Status: Completed | Type: Observational
Sponsor: Mann Eye Institute (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-24-01
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- TECNIS Odyssey IOL
  Interventions: Device: TECNIS Odyssey IOL

INTERVENTIONS:
Device: TECNIS Odyssey IOL — Implantation with the TECNIS Odyssey IOL

SUMMARY:
This study is a single center, ambispective study of visual outcomes after successful bilateral cataract surgery. Subjects will be assessed at least 3 months postoperatively at a single visit. Clinical evaluations will include administration of the AIOLIS and OSDI questionnaires, as well as measurement of visual acuities at distance, intermediate, and near.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged 50 years and older who underwent bilateral cataract surgery with Odyssey IOL implantation.

Exclusion Criteria:

* Significant ocular comorbidities (e.g., macular degeneration, glaucoma).
* < 2 weeks post YAG capsulotomy.
* Best corrected distance visual acuity worse than 20/25.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible test subjects will be aged 50 years and older who underwent bilateral cataract surgery with Odyssey IOL implantation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Visual Acuity at Distance (6m) logMAR | 3 months postoperative
  Photopic and mesopic, binocular and monocular, and uncorrected and distance corrected
Visual Acuity at Intermediate (66cm) logMAR | 3 months postoperative
  Photopic and mesopic, binocular and monocular, and uncorrected and distance corrected
Visual Acuity at Near (40cm) logMAR | 3 months postoperative
  Photopic and mesopic, binocular and monocular, and uncorrected and distance corrected
Visual Acuity at Near (33cm) logMAR | 3 months postoperative
  Photopic and mesopic, binocular and monocular, and uncorrected and distance corrected

SECONDARY OUTCOMES:
Assessment of IntraOcular Lens Implant Symptoms (AIOLIS) Questionniare | 3 months postoperative
  The AIOLIS has 37 questions about symptoms, perceptions of general vision, and frequency of wearing glasses or contact lenses. Lower scores for the symptom questions indicate lower frequency and both of visual disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Brunson, OD, Principal Investigator — Mann Eye Institute
Locations (1):
- Mann Eye Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No